CLINICAL TRIAL: NCT03205189
Title: Comparison Between Pre-operative Prescription Delivered During Anesthesia Consultation or Post-operative Prescription: a Randomized Prospective Trial
Brief Title: Comparison Between Pre-operative Prescription Delivered During Anesthesia Consultation or Post-operative Prescription
Acronym: AMBUPRESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015/119/SC
Record Dates: First submitted 2017-06-15; First posted 2017-07-02 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Postoperative Pain; Ambulatory Surgery; Anesthesia; Postoperative Complication
Keywords: postoperative pain; ambulatory surgery; general anesthesia; anesthesia consultation; post-op prescription
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: This is a randomized, prospective, study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-operative prescription group (Other): This group will have a pre-operative prescription delivered during the preoperative anesthesia clinic.
  Interventions: Other: Comparison between pre-operative prescription and post-operative prescription
- Postoperative prescription group (Other): This group will receive the postoperative prescription.
  Interventions: Other: Comparison between pre-operative prescription and post-operative prescription

INTERVENTIONS:
Other: Comparison between pre-operative prescription and post-operative prescription — The first group will have a pre-operative prescription delivered during the preoperative anesthesia clinic and the second group will receive the postoperative prescription.

SUMMARY:
This study evaluates the comparison of the incidence of postoperative home pain after ambulatory surgery with general anesthesia between a group with pre-surgical prescription delivered during anesthesia preoperative clinic and a group with postoperative prescription.

DETAILED DESCRIPTION:
The ambulatory surgery increased over the last twenty years in France. The management of home pain after ambulatory surgery is a major challenge because it is the principal complication after day surgery with several consequences: nausea and vomiting, chronic pain, functional impairment with handicap, sleeping troubles, extra-hospital consultation. Management of home pain remains currently could be performed in ambulatory surgery. The French Society of Anesthesiology recommends to deliver pre-surgical prescription during the preoperative anesthesia clinic but this guideline is not bases on evidence in the literature. Also, we have previously shown in a retrospective non-randomized work a decrease of postoperative home pain in patient with general anesthesia. The main objective of this controlled and comparative study is to compare the incidence of postoperative home pain after ambulatory surgery with general anesthesia between a group with pre-surgical prescription delivered during anesthesia consultation and a group with postoperative prescription.

ELIGIBILITY:
Inclusion Criteria:

* Any major ambulatory surgery patient with general anesthesia.

Exclusion Criteria:

* Pregnancy.
* Minor patient.
* ASA score > 3.
* lack of general anesthesia.
* General anesthesia combined with locoregional anesthesia.
* Contraindication to ambulatory surgery.
* Chronic pain.
* chronic analgesic consumption.
* no indication of non steroidal anti-inflammatory drug, paracetamol with codeine and morphine.
* Active or old drug addiction.
* Cognitive disorders or dementia.
* Serious psychiatric disorders.
* Patient under curatorship or tutorship.
* No social protection
* Misunderstanding of the French language
* Patient participating in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Early home pain after ambulatory surgery | 24 hours after ambulatory surgery
  The primary outcome is the incidence of at least one home pain experience with intensity greater than 3 on a scale from 0 to 10 within 24 hours after surgery.

SECONDARY OUTCOMES:
Intense painful experience during hospitalisation | Day 1
  Incidence of a pain experience at mobilization or at rest of intensity greater than 3 on a scale from 0 to 10 during hospitalisation.
Low painful experience during hospitalisation | Day 1
  Incidence of a pain experience at mobilization or at rest of intensity lower than 3 on a scale from 0 to 10 during hospitalisation.
Low home pain experience | 24 hours after ambulatory surgery
  Incidence of a pain experience at mobilization or at rest of intensity lower than 3 at home on a scale from 0 to 10 within 24 hours after surgery
Intense home pain experience | Within 7 days after ambulatory surgery
  Incidence of home pain at mobilization or at rest of intensity greater than 3 on a scale from 0 to 10 within 7 days after surgery.
Low home pain experience | Within 7 days after ambulatory surgery
  Incidence of home pain at mobilization or at rest of intensity lower than 3 at home on a scale from 0 to 10 within 7 days after surgery
Adherence to analgesic treatment | Within 7 days after ambulatory surgery
  Adherence to analgesic treatment in relation to prescription (yes or not)
Patient's satisfaction | Within 7 days after ambulatory surgery
  Patient's satisfaction with prescribed treatment (scale from 0 to 10, satisfying opinion defined by a score greater than 8)
Use of morphine analgesics | Within 7 days after ambulatory surgery
  Incidence of morphine analgesic use

CONTACTS AND LOCATIONS:
Overall Officials: Vincent COMPERE, Pr, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Selim J, Djerada Z, Chaventre C, Clavier T, Dureuil B, Besnier E, Compere V. Preoperative analgesic instruction and prescription reduces early home pain after outpatient surgery: a randomized controlled trial. Can J Anaesth. 2022 Aug;69(8):1033-1041. doi: 10.1007/s12630-021-02023-0. Epub 2021 May 13. PMID 33982238